CLINICAL TRIAL: NCT00148005
Title: Prevalence, Etiology and Therapy of Micturition Disorders of Children With a Mental and/or Motoric Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003/267
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Micturition Disorder
MeSH Terms: conditions — Urination Disorders | interventions — Surveys and Questionnaires; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Questionnaire and micturition and drinking diaries
Procedure: Clinical and functional examination (uroflowmetry, bladder scan and video-urodynamic examination)
Behavioral: Adaptation of the drinking scheme
Drug: Anticholinergic therapy
Behavioral: Micturition clock

SUMMARY:
Investigation of the prevalence etiology and therapy of micturition disorders of children with a mental and/or motoric disability

DETAILED DESCRIPTION:
Overview of the problem by a questionnaire, diary of micturition and drinking behaviour, filled out by the parents or by the staff of the institution.

Investigation of the etiology by clinical and functional examination (uroflowmetry, bladder scan, video-urodynamic examination).

Frequency:

* Uroflowmetry: two periods of two weeks, with 6 weeks break between both periods. During the follow-up period every 3 months during 12 months
* Bladder scan: once during the periods of the uroflowmetry
* Video-urodynamic examination: once in selected participants, after consent of the parents
* Adaptation of the drinking behaviour: start after two weeks of observation, after uroflowmetry and bladder scan. Continuous proces.
* Therapeutic measures (medication, miction clock): start after 10 weeks of observation or after video-urodynamic examination.

Development of a therapeutic plan: adaptation of the micturition and drinking behaviour, anticholinergic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children with a motoric and/or mental disability
* 4-14 years

Exclusion Criteria:

* Known neurogenic bladder disorder

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250
Dates: Start 2004-09

PRIMARY OUTCOMES:
Prevalence of micturition disorders
Etiology of micturition disorders after 10 weeks observation
Influence of drinking scheme on bladder capacity and micturition continence after 10 weeks observation

SECONDARY OUTCOMES:
Efficacy of the therapy after 3, 6, 9, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Erik Van Laecke, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be